CLINICAL TRIAL: NCT01857778
Title: Breast Tissue Before And After Breastfeeding Or The Use Of A Breast Pump
Status: Completed | Type: Observational
Sponsor: Foundation for Maternal Infant and Lactation Knowledge (Other)
Responsible Party: Principal Investigator, Nicole McDowell, Researcher, Foundation for Maternal Infant and Lactation Knowledge
Other Study IDs: 1990
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2011-10

CONDITIONS: To Collect Measurements of the Nipple; To Record Clinical Observations of the Nipple, Areola, and Breast Tissue Before and After Breastfeeding; To Record Clinical Observations of the Nipple, Areola, and Breast Tissue Before and After Expressing Milk With 3 Different Electric Breast Pumps.
Keywords: Breastfeeding; Breast tissue; Breast pump
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lactating Women

SUMMARY:
There will be breast tissue changes after use of a breast pump.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women who were breastfeeding.

Exclusion Criteria:

* Non breastfeeding or non lactating women.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Lactating women.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Breast Tissue Change | 10 minutes
  Lactating women used a 1 of 3 breast pumps or breastfed for 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jimi Francis, PhD, Principal Investigator — Foundation for M.I.L.K.
Locations (1):
- Renown Medical Center, Reno, Nevada, United States